CLINICAL TRIAL: NCT00100425
Title: Central Nervous System Modulation of Visceral Pain in Persian Gulf War Syndrome
Brief Title: Characterization of Pain Processing Mechanisms in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CADE-ARCD2
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Visceral Hypersensitivity; Visceral Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Visceral Pain

INTERVENTIONS:
Procedure: Viceral Perception Testing

SUMMARY:
The purpose of this study is to provide new information and to determine which kinds of brief, tolerable, experimental pain are affected by the drugs being studied in patients with irritable bowel syndrome, a disease that causes chronic abdominal pain. The effects of dextromethorphan, naloxone, and fentanyl on experimental pain stimuli will be tested in these studies to better understand what causes irritable bowel syndrome.

ELIGIBILITY:
* Patients with irritable bowel syndrome and healthy pain-free individuals (as controls) will be studied.
* No medical condition that would contraindicate use of dextromethorphan, fentanyl or naloxone.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- Malcolm Randall VA Medical Center, Gainesville, Florida, United States